CLINICAL TRIAL: NCT06549777
Title: Body-oriented Psychotherapy vs. Psychoeducation and Treatment Information for Individuals With a History of Child Maltreatment and Trauma-related Symptoms: Assessing Safety, Feasibility, Acceptability, and Preliminary Outcomes
Brief Title: Body-oriented Psychotherapy for Individuals With a History of Child Maltreatment and Trauma-related Symptoms
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Monique Pfaltz (Other)
Collaborators: Stockholm University (Other)
Responsible Party: Sponsor-Investigator, Monique Pfaltz, Professor, Mid Sweden University
Organization: Mid Sweden University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KPB-Study
Record Dates: First submitted 2024-08-05; First posted 2024-08-12 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Safety, Psychological; Acceptability of Health Care; Psychological Safety; Maltreatment, Child; Post Traumatic Stress Disorder; Complex Post-Traumatic Stress Disorder
Keywords: Safety; Feasibility; Body-oriented intervention; Somatic Experiencing; Psychological safety; Social safeness; Childhood maltreatment; Post traumatic stress disorder; Complex Post traumatic stress disorder; Interoception; Depression
MeSH Terms: conditions — Patient Acceptance of Health Care; Stress Disorders, Post-Traumatic; Depression

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to either an intervention group (receiving brief psychoeducation - reading a text which takes approximately 30 min to read - about PTSD/CPTSD, including information about how to seek help/treatment within the Swedish health care system + 15-session body-oriented SE treatment conducted over 20 weeks) or a control group (receiving the same psychoeducation and information about treatment possibilities + regular phone calls during the same period to provide updates on their well-being and if they started a treatment).
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SE-group (Experimental): The participant allocated to the SE-group will receive the same information sheet (taking approximately 30 minutes to read) as the control group in addition to the SE-treatment (Payne et al., 2010) consisting of 15 sessions conducted by certified SE therapists, with an adapted focus on specifically (C)PTSD and CM, as described in a manual available upon request from the authors. Sessions 1-3 focus on general practices for establishing a sense of self, contacting own space and positive interoceptive experiences. Sessions 4-6 aim to establish self-defensive behavior, to get into contact with one's own strength and with a sense of autonomy and attachment. Sessions 7-9 focus on working with depression, shame and anger. Sessions 10-12 include work with childhood patterns and sessions 13-15 aim at integrating the previous therapeutic work in daily life situations and at recapitulating some of the interventions.
  Interventions: Behavioral: SE-group
- Control (Active Comparator): The control group will receive an information sheet with psychoeducation about (C)PTSD (e.g., advice on self-care for symptom relief, available treatment options) and information about how to seek help/treatment within the Swedish health care system (taking approx.30 minutes to read). During the 20-week period the participant will be free to seek treatment of any kind and will additionally receive three phone calls (10 -15 minutes each time) from a research assistant (supervised by one of the project members). These calls aim to monitor participants' progress in seeking treatment and address any questions or concerns they may have regarding their involvement in the study. In addition, the calls aim to remind participants of completing the study questionnaires, in case they missed completing one or several of them.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: SE-group — Psychoeducation and information about treatment possibilities + SE-treatment
  Arms: SE-group
Behavioral: Control — Psychoeducation and information about treatment possibilities + Phone
  Arms: Control

SUMMARY:
This Pilot Randomized Controlled Trial (RCT) overall aim is to establish the safety, feasibility, acceptability and preliminary effects of a body-oriented psychotherapy, Somatic Experiencing (SE), on social functioning and mental health among adults with a history of Child Maltreatment (CM) and symptoms of posttraumatic stress disorder (PTSD) or complex posttraumatic stress disorder (CPTSD). Participants will be randomized either to an SE-group (n=25, psychoeducation, and information about treatment possibilities + 15-session SE treatment) or to a control group (n=25, same psychoeducation and information about treatment possibilities + regular phone calls to provide updates on their well-being and if they started a treatment). Given the lack of research on the effect of SE on Psychological Safety in this population, while SE has not yet been introduced into the Swedish health care system, special consideration will be given to participant safety, feasibility and acceptability of the SE-treatment. This includes monitoring (and assessing) for serious adverse events (SAEs) and adverse events (AEs), if conducting an RCT on SE in our target sample is feasible (e.g., achieving the target sample goal, assessing attrition rates and session attendance) and the acceptance of the used SE intervention (e.g., positive evaluations and willingness to recommend the treatment). Next to assessing safety, feasibility and acceptability, preliminary outcomes (self-report and experimental measures) will be evaluated at pre-treatment, post-treatment (20 weeks after pre), and at a 20-week follow-up, assessing primary outcomes (Psychological Safety) and secondary outcomes (Social Safeness, PTSD, CPTSD, Depression), as well as additional factors (e.g., interoception) that could contribute to decreased mental health and social functioning issues. Additionally, participants' behavioral (e.g., interpersonal distance) and physiological responses (HR, HRV, EDA) to social stimuli will be assessed pre- and post-treatment in an experimental setup to explore SE's potential to reduce Negative Affect and increase Positive Affect (Activated, Relaxed, Safe/Content) in response to social stress.

DETAILED DESCRIPTION:
Adults with a history of CM may struggle with psychological safety on both an emotional and physiological level, such as interpreting neutral facial expressions as negative/threatening or experiencing distress when approaching or being approached by others (Lüönd et al., 2022; Pfaltz et al., 2019). However, just as the social environment can be perceived as threatening, adults with CM-history can also experience absence of safety cues (e.g., perceived social support) which not only heightens the risk of developing and maintaining PTSD and CPTSD (Scott et al., 2023), but also impair social functioning further (cf. Pfaltz et al., 2022).

Although effective interventions like trauma-focused CBT exist for treating mental disorders such as PTSD (Lewis et al., 2020), they less often focus on facilitating feelings related to psychological safety such as social safeness (i.e., the extent to which individuals perceive their world as safe, warm, and soothing). This is problematic because exaggerated stress reactions and somatic symptoms may persist after treatment (Larsen et al., 2019) and social safeness could be a protective factor against these symptoms (Gilbert, 2020). Studies have e.g. shown that the presence of a friend can reduce stress reactions in individuals exposed to social stress (Heinrichs et al., 2003), and exposure to safety-related texts/images can reduce exaggerated stress responses to threatening situations (Gillath & Karantzas, 2019). Thus, social safeness may be crucial for regulating affective states.

Therefore, it is necessary to evaluate interventions that not only reduce symptoms of mental disorders but also actively focus on facilitating social, emotional, and body sensations related to feeling safe, particularly for individuals with CM-histories that not only suffer from mental disorders, but also lack protective factors that could inhibit it, such as caring support from others or self. One potential intervention is SE, a body-oriented approach (Levine, 1997). Unlike CBT and exposure-based interventions, SE focuses more on interoception and musculoskeletal sensations rather than primary focus on cognitions to promote affective self-regulation and resilience to stress (Payne, 2015). Through SE, clients are assumed to learn to manage unpleasant emotions and reduce negative bodily reactions, while identifying positive bodily sensations that provide safety and calmness. This might help clients to be present in their surroundings and potentially restore their ability to feel socially safe both physically and psychologically.

Preliminary results from our own (to be published) studies show that SE has a short-term effect (one session) on increased perceived psychological safety in adults with a history of CM compared to a control group. Systematic reviews and meta-analyses have as well indicated that SE can reduce symptoms of PTSD, depression, and somatic symptoms (Heim et al., 2023; Kuhfuß et al., 2021). However, there is a research gap concerning the feasibility, acceptability and preliminary long-term effects of SE on facilitating psychological safety in individuals with a history of CM and PTSD/CPTSD symptoms.

Accordingly, we will conduct a pilot RCT, adhering to the Consolidated Standards of Reporting Trials (Schulz, 2010), to evaluate the feasibility of SE, acceptability, and safety as well as to explore the potential of SE (preliminary outcomes) for improving social functioning and mental health for adult participants with a CM-history and symptoms of (C)PTSD. Participants meeting these criteria will be randomly allocated to either an SE-group (n=25) or to a control group (n=25). Self-report measures will be collected pre, post-treatment, and at a 20-week FU assessing primary outcomes (Psychological Safety) and secondary outcomes (Social Safeness, PTSD, CPTSD, Depression, Sense of Disrupted Body Boundaries, Interoceptive Awareness, Attachment style, Social Support, and Somatic symptoms). Potential influencing variables (Socio-Demographics, Attitudes towards Psychotherapy, CM history, Attachment style, Interoceptive Awareness, Social Phobia, and Therapeutic Alliance) will be analyzed to explore potential mechanisms of treatment responses in primary and secondary outcomes. Moreover, participants will attend a physical visit (experimental study part) at Stockholm University (SU) where we assess behavioral (e.g., interpersonal distance), physiological responses (HR, HRV and EDA) and affective responses (e.g., negative affect) to social stimuli (e.g., facial expressions).

In addition to primarily assessing safety, feasibility and acceptability of the intervention (See brief summary), we will test the following hypotheses regarding preliminary effects of the intervention:

Primary hypothesis (Primary outcomes):

1. Participants in the SE-group, compared to the control group, will show higher levels of Psychological Safety at post-treatment and FU.

   Secondary hypothesis (Secondary outcomes):
2. Participants in the SE-group, compared to the control group, will show higher levels of Social Safeness at post-treatment and FU.
3. Participants in the SE-group, compared to the control group, will show lower levels of PTSD, CPTSD, Depression, Sense of Disrupted Body Boundaries and Somatic Symptoms at post-treatment and FU.
4. Participants in the SE-group, compared to the control group, will show higher levels of Attachment Security, Interoceptive Awareness, and Social Support at post-treatment and FU. 5. Based on preliminary results from our short-term intervention study, higher levels of CM will predict a stronger treatment response, indicated by a stronger increase in Psychological Safety in the SE-group compared to the control group.

Hypotheses related to the experimental study part:

6. Participants in the SE-group, compared to the control group, will rate neutral facial expressions less negatively from pre- to post-treatment.

7. Participants in the SE-group, compared to the control group, will show greater decrease in preferred interpersonal distance from pre- to post-treatment.

8. Participants in the SE-group, compared to the control group, will show improved affective/physiological self-regulation (self-reports on TPAS, body sensations, higher HRV, lower HR, and decreased EDA response) following exposure to attachment primes (recalling and visualization interpersonal insecure and secure attachment-related experiences) from pre- to post-treatment.

Method

To characterize the sample (presence of mental disorders) and to assess exclusion criteria we will employ sections of the MINI (Sheehan et al., 1998) that is relevant for our study population.

Before randomization, participants will complete four experimental paradigms at SU, including: "stop-distance task," (measuring participants' preferred physical distance towards strangers, see Lüönd et al., 2022) and a "rope exercise" measuring safety within one's personal space (for exploratory purposes). Then, the participants' physiological (HR, HRV, EDA) and self-reported responses to facial expressions (Pfaltz et al., 2019) will be assessed. Lastly, the participants' affective (self-reported) and physiological (HR, HRV, EDA) self-regulation in response to attachment primes (described above) will be evaluated. After the physical visit, randomization to SE or control will take place.

Adverse events (AEs) will be defined as any unfavorable medical occurrences or undesirable experiences (e.g., suicidal thoughts, dependency, symptom worsening, hopelessness, failure, stigma, quality of treatment) encountered by participants during the study-period, regardless of their relation to the study.

All participants will complete symptom scales (ITQ and PHQ9) at pre, repeatedly during, post and at FU. A symptom increases on ITQ from pre to any of the follow-up measurement points of 50% - 79% is considered an AE, an increase of 80% or more is considered a SAE. If participants score ≥ 1 on suicidality item 9 (PHQ-9) at any of the measurement points, we will conduct a risk assessment and based on this determine if one of the following applies: (i) death by suicide; (ii) suicide attempt; (iii) suicidal crisis without attempt; (iv) self-harming behaviors and thoughts of self-harm.

(i) - (iv) are counted as SAE if they:

1. result in death and/or:
2. are life-threatening
3. require hospitalization or prolongation of existing hospitalization
4. result in significant disability or incapacity Thoughts and behaviors that do not result in a), b), c), or d) will be considered AE.

Determination of whether an (S)AEs is related to the SE-treatment will be based on whether the event is unexpected or unexplained given participants' clinical development, previous medical conditions, medications or interventions. An AE form will be provided to therapists for completion at the end of each session, instructed to report AEs within 24 hours and SAEs directly to the research team, who will review (and consult with a psychiatrist in the project) and assess the nature of each event(s) to decide on appropriate actions such as potential participant withdrawal of the study.

At post-treatment, AEs will be assessed using the NEQ. Feasibility and acceptability will be evaluated via participant-written evaluations, analyzed both quantitatively (e.g., percent of satisfactory with SE and recommend SE to others) and qualitatively (e.g., thematic analysis). All SE sessions will be audio-recorded for exploratory analysis and to assess treatment integrity and fidelity. A random selection of sessions will be independently scored, by an independent assessor, for fidelity to ensure adherence to the treatment manual.

There are no efficacy studies on longitudinal interventions for Psychological Safety, to enable adequate a priori power calculations and resource constraints allowing for a sample size (approximately n=25 in each group), our study will follow Lakens (2022) recommendations: assessing precision via confidence interval widths and explore detectable effect sizes across various power levels via sensitivity power analysis. Based on the outcome, the BUCSS R package (See Anderson et al., 2017) for implementing Bias- and Uncertainty-Corrected Sample Size, a method of correcting for publication bias and uncertainty when planning sample sizes in a future study from an original study.

Analyses will follow an intention-to-treat approach, including all randomized participants, even those who do not complete the study. For primary and secondary outcomes, we plan to use linear mixed models to handle missing data, assuming data are missing at random. Time (pre, post, treatment, and FU) and Group (SE vs. control) will be fixed effects, with participants as random effects. Treatment efficacy will be indicated by a significant time-by-treatment interaction. Potential moderators influencing treatment effects will be analyzed as covariates in the mixed model analysis. Clinically significant changes in (C)PTSD and Depression scores will be analyzed by calculating a Reliable Change Index (RCI), classified as "improved," "worsened," or "unchanged" based on changes in symptom scores exceeding relevant RCI values (See Cloitre et al. 2021). Behavioral and physiological responses at the experimental study part will be analyzed using a similar analytic approach (linear mixed models) or ANOVA. HRV measurement will include both common frequency estimates (e.g., HF) and time domain estimates (e.g., rMSSD).

Outliers will be identified using univariate and multivariate detection methods, such as Cook's distance (with values >1 indicating an outlier) and standardized residuals (±3.29 indicating an outlier, Tabachnick & Fidell, 2013). If outliers are identified, we aim to present results both with outliers, and with the adjustment for outliers, and/or consider using robust maximum likelihood (MLR) estimation, which is more robust against outliers.

ELIGIBILITY:
Inclusion Criteria:

* Adults (18 years or older).
* Proficiency in Swedish Language.
* Access to a computer/internet.
* Meeting CTQ-cutoff for CM history (CTQ rating higher than 'none / minimal' in at least one of the subscales according to Bernstein and Fink (1998) (i.e. ≥10 for emotional neglect, ≥ 8 for physical neglect, ≥9 for emotional abuse, ≥8 for physical abuse and ≥6 for sexual abuse).
* Meeting at least moderate/severe PTSD or complex PTSD symptoms on the ITQ.
* If taking medication, it must have been ongoing for at least 3 months and the dose must have been stable for 1 month.
* Signed informed consent provided.

Exclusion Criteria:

* Participants screen positive for alcohol (AUDIT) or substance abuse (DUDIT).
* Psychotic symptoms, ongoing manic episode, acute suicidality.
* If ongoing medication has an impact on the physiological data (ECG) recorded during the social paradigms, physiological data will be excluded from the analyses (but not exclusion for the treatment).
* Have current (pre-assessment) ongoing psychological treatment focusing on social safeness, PTSD or complex PTSD.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-09-06 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
The Neuroception of Psychological Safety Scale (NPSS; Morton et al., 2024) | Pre-treatment, post-treatment (20 weeks after pre-treatment) and follow-up (20-week after post-treatment).
  To measure psychological safety the 29-item NPSS will be used, which covers social engagement, compassion, and body sensations related to feeling safe. Items on NPSS are scored on a Likert scale ranging from 1 (strongly disagree) to 5 (strongly agree) the extent to which participants agree with the items (e.g., "My body felt relaxed") higher total score indicates higher feelings of psychological safety.

SECONDARY OUTCOMES:
Social Safeness and Pleasure Scale Scale (SSPS; Gilbert et al., 2009; Isaksson et al, 2022) | Pre-treatment, post-treatment (20 weeks after pre-treatment) and follow-up (20-week after post-treatment).
  To measure Social Safeness (a state related to feeling psychological safe) the 11- item SPSS will be used. Items are scored on a Likert scale ranging from 1 (almost never) to 5 (almost all the time) to measure the extent to which participants agree with the items (e.g., "I feel easily soothed by those around me."). Scores are added together to produce a total score in the range 11-55, with higher scores representing higher perceived social safeness.
International Trauma Questionnaire (ITQ; Cloitre et al., 2018) | Pre-treatment, during treatment post-treatment (20 weeks after pre-treatment) and follow-up (20-week after post-treatment).
  To measure PTSD and CPTSD the 18-item ITQ will be used. Participants will indicate on a Likert scale ranging from 0 (Not at all) to 4 (Extremely) the extent to which they agree with the items (e.g., "Having upsetting dreams that replay part of the experience or are clearly related to the experience?"). Probable PTSD is considered when at least one symptom from all PTSD symptom clusters and at least one PTSD-related functional impairment has a score ≥2. Probable complex PTSD is confirmed if all PTSD criteria are met, and at least one symptom in each DSO cluster (Disorders in self-organization) and at least one DSO-related functional impairment are ≥2.A symptom increases on ITQ from pre to any of the follow-up measurement points of 50% - 79% is considered an AE, an increase of 80% or more is considered a SAE.
The Patient Health Questionnaire (PHQ-9; Kroenke et al., 2001) | Pre-treatment, during treatment, post-treatment (20 weeks after pre-treatment) and follow-up (20-week after post-treatment).
  The PHQ-9 (Korienke et al., 2001) is a 9-item questionnaire measuring depressive symptoms and suicidal ideations. Participants will indicate on a Likert scale ranging from several days (0) to nearly every day (3) the extent to which they agree with the items (e.g., "Little interest or pleasure in doing things."). High scores indicate a higher frequency of depressive symptoms over the past two weeks. We will consider a participant to have suicidal ideations if they score 1 or > on item 9 "Thoughts that you would be better off dead or of hurting yourself in someway".
The Body Boundaries Survey (BBS; Krzewska & Dolińska- Zygmunt, 2013) | Pre-treatment, post-treatment (20 weeks after pre-treatment) and follow-up (20-week after post-treatment).
  To measure sense of disrupted body boundaries the 17 item BBS will be used. Participants will indicate on a Likert-scale ranging from 1 (Definitely don't agree) to 5 (Strongly agree) the extent to which they agree with items (e.g., "When someone gets too close to me, I feel as if he/she is invading my physical space."). Higher scores indicated a stronger sense of disrupted body boundaries
The Multidimensional Assessment of Interoceptive Awareness (MAIA-2; Mehling et al., 2018). | Pre-treatment, during treatment, post-treatment (20 weeks after pre-treatment) and follow-up (20-week after post-treatment).
  To measure interoceptive awareness three subscales (Self-Regulation, Noticing, Trusting and Emotional awareness), i.e., 16-items from the MAIA-2 will be used (based on results from our unpublished study). Participants will indicate on a Likert scale ranging from 1 (Never) to 5 (Always) the extent to which they agree with each item (e.g., "I can return awareness to my body if I am distracted."). Higher scores indicate stronger interoceptive awareness.
Experiences in close relationships (ECR-RS; Brennan et al., 1998; Sarling et al., 2021) | Pre-treatment, post-treatment (20 weeks after pre-treatment) and follow-up (20-week after post-treatment).
  To measure adult attachment style, the 9-item ECR-12 will be used. Participants will indicate on a Likert scale ranging from 1 (Strongly disagree) to 7 (strongly agree) the extent to which they agree with the items (e.g., "I worry about being abandoned by the person closest to me."). Low scores indicate a perceived secure attachment, and high scores indicate a perceived insecure attachment.
The multidimensional scale of perceived social support (MSPSS; Zimet et al., 1988; Ekbäck et al., 2013) | Pre-treatment, post-treatment (20 weeks after pre-treatment) and follow-up (20-week after post-treatment).
  To measure perceived social support the 12-item MSPSS will be used. Participants will indicate on a Likert scale ranging from 1 (very strongly disagree) to 7 (very strongly agree) the extent to which they agree with each item (e.g., "I get the emotional help and support I need from my family.").
The Patient Health Questionnaire-15 (PHQ-15; Korienke et al., 2002) | Pre-treatment, post-treatment (20 weeks after pre-treatment) and follow-up (20-week after post-treatment).
  To measure somatic symptoms the 15 item PHQ-15 will be used. Participants will indicate on a Likert-scale ranging from 1 (not bothered at all) to 3 (bothered a lot)" to the extend they have been bothered by symptoms during the past four weeks (e.g., "Stomach pain."). Total scores range from 0-30 (for women), 0-28 (men), with scores of ≥5, ≥10, ≥15 representing mild, moderate and severe levels of somatization.

OTHER OUTCOMES:
Childhood Trauma Questionnaire-Short Form (CTQ-SF; Bernstein et al., 2003; Gerdner & Allgulander, 2009) | Pre-treatment
  To measure CM histories, the 28-item CTQ-SF will be used. Participants will indicate on a Likert scale ranging from 1 (Never true) to 5 (Always true) the extent to which they agree with the items (e.g., "I believe I was emotionally abused."). Higher total score indicates more exposure to CM. To be included in the study the participants need to reach cut-off scores categorized as higher than 'none / minimal' in at least one of the subscales according to Bernstein and Fink (1998) (i.e. ≥10 for emotional neglect, ≥ 8 for physical neglect, ≥9 for emotional abuse, ≥8 for physical abuse and ≥6 for sexual abuse).
Life event-checklist (LEC-5; Weathers et al., 2013) | Pre-treatment
  To assess participant's trauma history, they will be asked to consider their entire lifespan and to indicate which out of 17 traumatic events have happened to themselves or to others (observed by the participant).
The Mini social phobia inventory (mini-SPIN; Connor et al., 2001) | Pre-treatment, post-treatment (20 weeks after pre-treatment) and follow-up (20-week after post-treatment).
  To measure symptoms of social phobia the 3-item mini-SPIN will be used. Participants will indicate on a 4-point Likert scale (0 = not at all; 4= extremely) the extent to which they agree with items (e.g., " I avoid activities in which I am the center of attention."). Higher scores indicate higher levels of social phobia.
The Working Alliance Inventory (WAI-S; Horvath, & Greenberg, 1989) | Post-treatment (20 weeks after pre-treatment)
  To measure the quality of the alliance (between therapist and participant) and study its relationship to treatment outcomes the 12-item WAI-S will be used. Participants and therapist will indicate on a 7-point Likert scale (1= never; 7 = always) the extent to which they agree how often items apply to them (e.g., "My therapist and I work towards common goals.". A higher score indicates a higher degree of working alliance.
Vividness and clarity of visualization (Mikulincer & Shaver, 2001) | Pre-treatment and post-treatment (20 weeks after pre-treatment)
  This scale is used exclusively during the experimental study-part.To assess vividness and clarity and emotionally of visualization during guided imagination task (after exposure to insecure and secure attachment primes), participants will rate the vividness and clarity of their visualization and how emotionally it was-on sliding scale ranging from 0 (not at all) to 100 (very much).
The Swedish version of the types of positive affect scale (TPAS; Gilbert et al., 2008; Lehmivaara et al., 2024, in press) | Pre-treatment and post-treatment (20 weeks after pre-treatment)
  This scale is used exclusively during the experimental study-part. To measure different types of state positive affect related to psychological safety before and after exposure to insecure and secure attachment primes, the 18-item TPAS will be used. Participants will indicate on a Likert scale ranging from 1 (not at all) to 5 (very much) the extent to which they agree with affective states in the present moment: Activated PA (e.g., excitement), Relaxed PA (e.g., calm). and Safe/Content PA (e.g., safe). Higher scores on each subscale indicated higher levels of currently experienced PA.
The Positive and Negative Affect Schedule Short form (PANAS-SF; Garcia,Nima & Lindskär, 2016; Watson, Clark, & Tellegen, 1988) | Pre-treatment and post-treatment (20 weeks after pre-treatment)
  This scale is used exclusively during the experimental study-part. To measure state negative affect before and after exposure to insecure and secure attachment primes, 5 items (affective states, e.g., "upset") from the PANAS-SF will be used. Participants will indicate on a Likert-scale ranging from 1 (very slightly) to 5 (very much) the extent to which they experience with affective states in the present moment (e.g., shame). Higher scores indicate a stronger current negative affective state.
The Subscale Body sensations on the The Neuroception of Psychological Safety (NPSS; Morton et al., 2022) | Pre-treatment and post-treatment (20 weeks after pre-treatment)
  This scale is used exclusively during the experimental study-part. To measure bodily sensations related to perceived safety before and after exposure to insecure and secure attachment primes, the 8-item subscale body sensation from NPSS will be used. Participants will indicate on a Likert scale ranging from 1 (strongly disagree) to 5 (strongly agree) the extent to which they agree with the items (e.g., "My body feels relaxed.").
Occurrence of Adverse events on the Negative Effects Questionnaire (NEQ; Rozental et al., 2016) | Post-treatment (20 weeks after pre-treatment assessment)
  To measure occurrence and characteristics of negative effects (AEs) in psychological treatments the 20-item NEQ will be used. The participants will indicate how they experienced and felt during the treatment with Yes or No to items such as "I felt more stressed" and if yes, they will indicate on 5-point Likert scale to what extent to which it was negative (1 = not at all; 5= extremely) and related to the treatment or not. We will consider a participant to have suicidal ideations if they score Yes on item 10.
Feasibility and acceptability of the SE-intervention and psychoeducation on surveys developed for this study | Post-treatment (20-weeks after pre-treatment) and Follow-up (20-week after post-treatment).
  To measure feasibility and acceptability, participants will indicate, how they subjectively experienced and felt during the study (e.g., experience of the intervention/partaking in the study as controls, positive and negative aspects of the treatment, the impact on their wellbeing, and be asked to offer suggestions for improvement), with both yes/no and open questions. Percentage of participants completing SE-treatment and completing outcome measures at the end of treatment and at FU will be calculated as well.
Alcohol Use Disorders Identification Test (AUDIT; Babor et al., 1989; Bergman & Kaellmen, 2002) | Pre-treatment (before inclusion to the study)
  To screen for alcohol misuse, we will use the 10 item AUDIT. Participants will indicate on a Likert scale ranging from (1) never to (5) daily on items (e.g., "How often do you drink six or more of such 'glasses' on a single occasion?").
Drug Use Disorders Identification Test (DUDIT; (Berman et al., 2005) | Pre-treatment (before inclusion to the study)
  To screen for drug misuse, us we will use the 10-item DUDIT. Participant will indicate on a scale ranging from never (1) to 4 times/week or more nearly every day (5) the extent to which they agree with the items (e.g., "How often do you use drugs other than alcohol? (Refer to the drug list on the back.)". If participant score 6 point or above (men) and 2 and above (women) indicate a problem with substance misuse can be present or has been present.
Ongoing medication, psychological treatment, and stable dosage | Pre-treatment (before inclusion to the study), during, Post-treatment (20-weeks after pre-treatment) and at Follow-up (20-week after post-treatment).
  To screen for ongoing medication or psychological treatment and stable dosage both before and during the study, 3 items developed for this study will be used. Participants will indicate with "Yes" or "No" to questions about whether their medication has been ongoing for three months prior to study inclusion, whether the dosage has been stable for at least one month, and whether they are currently undergoing psychological treatment for social safeness, PTSD, or CPTSD. Throughout the study, participants will also be asked regularly if there have been any changes in medication or if they have attended other psychological treatments and be asked to provide open answer to why.

CONTACTS AND LOCATIONS:
Overall Officials: Monique Pfaltz, Principal Investigator — +46101428300
Locations (1):
- Mid Sweden university and Stockholm university, Stockholm, Stockholm County, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Anderson SF, Kelley K, Maxwell SE. Sample-Size Planning for More Accurate Statistical Power: A Method Adjusting Sample Effect Sizes for Publication Bias and Uncertainty. Psychol Sci. 2017 Nov;28(11):1547-1562. doi: 10.1177/0956797617723724. Epub 2017 Sep 13. PMID 28902575
- [Background] Berman AH, Bergman H, Palmstierna T, Schlyter F. Evaluation of the Drug Use Disorders Identification Test (DUDIT) in criminal justice and detoxification settings and in a Swedish population sample. Eur Addict Res. 2005;11(1):22-31. doi: 10.1159/000081413. PMID 15608468
- [Background] Bernstein DP, Stein JA, Newcomb MD, Walker E, Pogge D, Ahluvalia T, Stokes J, Handelsman L, Medrano M, Desmond D, Zule W. Development and validation of a brief screening version of the Childhood Trauma Questionnaire. Child Abuse Negl. 2003 Feb;27(2):169-90. doi: 10.1016/s0145-2134(02)00541-0. PMID 12615092
- [Background] Bergman H, Kallmen H. Alcohol use among Swedes and a psychometric evaluation of the alcohol use disorders identification test. Alcohol Alcohol. 2002 May-Jun;37(3):245-51. doi: 10.1093/alcalc/37.3.245. PMID 12003912
- [Background] Cloitre M, Shevlin M, Brewin CR, Bisson JI, Roberts NP, Maercker A, Karatzias T, Hyland P. The International Trauma Questionnaire: development of a self-report measure of ICD-11 PTSD and complex PTSD. Acta Psychiatr Scand. 2018 Dec;138(6):536-546. doi: 10.1111/acps.12956. Epub 2018 Sep 3. PMID 30178492
- [Background] Cloitre M, Hyland P, Prins A, Shevlin M. The international trauma questionnaire (ITQ) measures reliable and clinically significant treatment-related change in PTSD and complex PTSD. Eur J Psychotraumatol. 2021 Jun 22;12(1):1930961. doi: 10.1080/20008198.2021.1930961. PMID 34211640
- [Background] Connor KM, Kobak KA, Churchill LE, Katzelnick D, Davidson JR. Mini-SPIN: A brief screening assessment for generalized social anxiety disorder. Depress Anxiety. 2001;14(2):137-40. doi: 10.1002/da.1055. PMID 11668666
- [Background] Ekback M, Benzein E, Lindberg M, Arestedt K. The Swedish version of the multidimensional scale of perceived social support (MSPSS)--a psychometric evaluation study in women with hirsutism and nursing students. Health Qual Life Outcomes. 2013 Oct 10;11:168. doi: 10.1186/1477-7525-11-168. PMID 24112950
- [Background] Gerdner A, Allgulander C. Psychometric properties of the Swedish version of the Childhood Trauma Questionnaire-Short Form (CTQ-SF). Nord J Psychiatry. 2009;63(2):160-70. doi: 10.1080/08039480802514366. PMID 19021077
- [Background] Gilbert P. Compassion: From Its Evolution to a Psychotherapy. Front Psychol. 2020 Dec 9;11:586161. doi: 10.3389/fpsyg.2020.586161. eCollection 2020. PMID 33362650
- [Background] Gillath O, Karantzas G. Attachment security priming: a systematic review. Curr Opin Psychol. 2019 Feb;25:86-95. doi: 10.1016/j.copsyc.2018.03.001. Epub 2018 Mar 15. PMID 29621693
- [Background] Heinrichs M, Baumgartner T, Kirschbaum C, Ehlert U. Social support and oxytocin interact to suppress cortisol and subjective responses to psychosocial stress. Biol Psychiatry. 2003 Dec 15;54(12):1389-98. doi: 10.1016/s0006-3223(03)00465-7. PMID 14675803
- [Background] Heim N, Bobou M, Tanzer M, Jenkinson PM, Steinert C, Fotopoulou A. Psychological interventions for interoception in mental health disorders: A systematic review of randomized-controlled trials. Psychiatry Clin Neurosci. 2023 Oct;77(10):530-540. doi: 10.1111/pcn.13576. Epub 2023 Aug 9. PMID 37421414
- [Background] Isaksson M, Holmbom Goh M, Ramklint M, Wolf-Arehult M. The Social Safeness and Pleasure Scale (SSPS): a psychometric evaluation of the Swedish version in a non-clinical sample and two clinical samples with eating disorders or borderline personality disorder. BMC Psychol. 2022 Dec 16;10(1):311. doi: 10.1186/s40359-022-01020-2. PMID 36527142
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-15: validity of a new measure for evaluating the severity of somatic symptoms. Psychosom Med. 2002 Mar-Apr;64(2):258-66. doi: 10.1097/00006842-200203000-00008. PMID 11914441
- [Background] Kuhfuss M, Maldei T, Hetmanek A, Baumann N. Somatic experiencing - effectiveness and key factors of a body-oriented trauma therapy: a scoping literature review. Eur J Psychotraumatol. 2021 Jul 12;12(1):1929023. doi: 10.1080/20008198.2021.1929023. eCollection 2021. PMID 34290845
- [Background] Larsen SE, Fleming CJE, Resick PA. Residual symptoms following empirically supported treatment for PTSD. Psychol Trauma. 2019 Feb;11(2):207-215. doi: 10.1037/tra0000384. Epub 2018 Jul 2. PMID 29963892
- [Background] Lewis C, Roberts NP, Gibson S, Bisson JI. Dropout from psychological therapies for post-traumatic stress disorder (PTSD) in adults: systematic review and meta-analysis. Eur J Psychotraumatol. 2020 Mar 9;11(1):1709709. doi: 10.1080/20008198.2019.1709709. eCollection 2020. PMID 32284816
- [Background] Luond AM, Wolfensberger L, Wingenbach TSH, Schnyder U, Weilenmann S, Pfaltz MC. Don't get too close to me: depressed and non-depressed survivors of child maltreatment prefer larger comfortable interpersonal distances towards strangers. Eur J Psychotraumatol. 2022 May 30;13(1):2066457. doi: 10.1080/20008198.2022.2066457. eCollection 2022. PMID 35957629
- [Background] Mehling WE, Acree M, Stewart A, Silas J, Jones A. The Multidimensional Assessment of Interoceptive Awareness, Version 2 (MAIA-2). PLoS One. 2018 Dec 4;13(12):e0208034. doi: 10.1371/journal.pone.0208034. eCollection 2018. PMID 30513087
- [Background] Mikulincer M, Shaver PR. Attachment theory and intergroup bias: evidence that priming the secure base schema attenuates negative reactions to out-groups. J Pers Soc Psychol. 2001 Jul;81(1):97-115. PMID 11474729
- [Background] Morton L, Cogan N, Kolacz J, Calderwood C, Nikolic M, Bacon T, Pathe E, Williams D, Porges SW. A new measure of feeling safe: Developing psychometric properties of the Neuroception of Psychological Safety Scale (NPSS). Psychol Trauma. 2024 May;16(4):701-708. doi: 10.1037/tra0001313. Epub 2022 Jul 18. PMID 35849369
- [Background] Payne P, Levine PA, Crane-Godreau MA. Somatic experiencing: using interoception and proprioception as core elements of trauma therapy. Front Psychol. 2015 Feb 4;6:93. doi: 10.3389/fpsyg.2015.00093. eCollection 2015. PMID 25699005
- [Background] Pfaltz MC, Passardi S, Auschra B, Fares-Otero NE, Schnyder U, Peyk P. Are you angry at me? Negative interpretations of neutral facial expressions are linked to child maltreatment but not to posttraumatic stress disorder. Eur J Psychotraumatol. 2019 Nov 11;10(1):1682929. doi: 10.1080/20008198.2019.1682929. eCollection 2019. PMID 31762947
- [Background] Pfaltz MC, Halligan SL, Haim-Nachum S, Sopp MR, Ahs F, Bachem R, Bartoli E, Belete H, Belete T, Berzengi A, Dukes D, Essadek A, Iqbal N, Jobson L, Langevin R, Levy-Gigi E, Luond AM, Martin-Soelch C, Michael T, Oe M, Olff M, Ceylan D, Raghavan V, Ramakrishnan M, Sar V, Spies G, Wadji DL, Wamser-Nanney R, Fares-Otero NE, Schnyder U, Seedat S. Social Functioning in Individuals Affected by Childhood Maltreatment: Establishing a Research Agenda to Inform Interventions. Psychother Psychosom. 2022;91(4):238-251. doi: 10.1159/000523667. Epub 2022 Apr 5. PMID 35381589
- [Background] Rozental A, Kottorp A, Boettcher J, Andersson G, Carlbring P. Negative Effects of Psychological Treatments: An Exploratory Factor Analysis of the Negative Effects Questionnaire for Monitoring and Reporting Adverse and Unwanted Events. PLoS One. 2016 Jun 22;11(6):e0157503. doi: 10.1371/journal.pone.0157503. eCollection 2016. PMID 27331907
- [Background] Schulz KF, Altman DG, Moher D; CONSORT Group. CONSORT 2010 Statement: updated guidelines for reporting parallel group randomised trials. BMC Med. 2010 Mar 24;8:18. doi: 10.1186/1741-7015-8-18. PMID 20334633
- [Background] Scott JG, Malacova E, Mathews B, Haslam DM, Pacella R, Higgins DJ, Meinck F, Dunne MP, Finkelhor D, Erskine HE, Lawrence DM, Thomas HJ. The association between child maltreatment and mental disorders in the Australian Child Maltreatment Study. Med J Aust. 2023 Apr 3;218 Suppl 6(Suppl 6):S26-S33. doi: 10.5694/mja2.51870. PMID 37004186
- [Background] Sheehan DV, Lecrubier Y, Sheehan KH, Amorim P, Janavs J, Weiller E, Hergueta T, Baker R, Dunbar GC. The Mini-International Neuropsychiatric Interview (M.I.N.I.): the development and validation of a structured diagnostic psychiatric interview for DSM-IV and ICD-10. J Clin Psychiatry. 1998;59 Suppl 20:22-33;quiz 34-57. PMID 9881538
- [Background] Watson D, Clark LA, Tellegen A. Development and validation of brief measures of positive and negative affect: the PANAS scales. J Pers Soc Psychol. 1988 Jun;54(6):1063-70. doi: 10.1037//0022-3514.54.6.1063. PMID 3397865